CLINICAL TRIAL: NCT02809989
Title: Multicentre, Prospective, Open, Non-interventional Study to Evaluate the Effect of Ovaleap® on the Pregnancy Rate and Clinical Effects as Well as the User-friendliness of the Ovaleap®-Pen in the Clinical Routine of the IVF- / ICSI-treatment.
Brief Title: A Study to Evaluate the Effect of Ovaleap® on the Pregnancy Rate and Clinical Effects as Well as the User-friendliness of the Ovaleap®-Pen.
Status: Completed | Type: Observational
Sponsor: Teva Pharma GmbH (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Other Study IDs: XM17-WH-40103
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Pregnancy Rate; Oocytes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ovaleap®: Single group prospective treatment cohort
  Interventions: Drug: Ovaleap®

INTERVENTIONS:
Drug: Ovaleap® — About 6-8 weeks of observation per patient from start of the stimulation therapy with Ovaleap® depending on the duration of the required stimulating therapy. Up to 10-11 months per patient for follow-up but only if in case of songraphically intact intrauterine pregnancy to determinate the "Baby-Take-Home-Rate" (live-births).

SUMMARY:
The aim of this non-interventional study is to extend the knowledge on effectiveness of Ovaleap® (number of oocytes and pregnancy rate) during routine IVF- or ICSI-treatment using a Gonadotropin-releasing hormone (GnRH) antagonist protocol in a large number of patients.

ELIGIBILITY:
Inclusion Criteria:

* Women with a medical indication for an ovarian stimulation therapy for the purposes of an IVF or ICSI.
* First-time ovarian stimulating therapy for an IVF or ICSI.
* Ovarian stimulation therapy exclusively with Ovaleap®.
* GnRH antagonist protocol.
* Body-Mass-Index (BMI) < 30 kg/m2.
* Duration of menstrual cycle 24 - 35 days.

  * Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* Combined application of IVF and ICSI
* Ovarian hyperstimulation with Ovaleap® with a consecutive "social freezing".
* Polycystic ovary syndrome (PCOS).
* Endometriosis (AFS (American Fertility Society) grade 3 and 4).
* Uterine myoma (intramural > 4 cm, submucosal).
* Hydrosalpinx (on one side or both sides).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who get an ovarian stimulation therapy with Ovaleap® as preparation for a technique of an assisted reproduction (here: In-vitro-Fertilisation (IVF) or Intracytoplasmatic Sperm Injection (ICSI).
Sampling Method: Non-Probability Sample
Enrollment: 507 (Actual)
Dates: Start 2016-03-31 (Actual); Primary Completion 2017-07-21 (Actual); Study Completion 2018-03-13 (Actual)

PRIMARY OUTCOMES:
Number of retrieved oocytes after ovarian stimulation therapy | 12 months
Clinical pregnancy rate | 12 months

SECONDARY OUTCOMES:
Number of days with administration of Ovaleap® | 12 months
Administered total dose of Ovaleap® | 12 months
Level of serum estradiol at the time of the last examination prior to induction of ovulation | 12 months
Endometrial thickness (mm) at time of the last sonography prior to induction of ovulation | 12 months
Used drugs for induction of the ovulation (recombinant Human chorionic gonadotropin (HCG), urinary HCG, GnRH agonist) | 12 months
Number of Metaphase II (MII)-oocytes | 12 months
Percentage fertilisation rate | 12 months
  * IVF: number of fertilised oocytes in 2-pro nucleus (2-PN)-stage / number of inseminated MII-oocytes as a percentage.
  * ICSI: number of fertilised oocytes in 2-PN-stage / number of injected MII-oocytes as a percentage.
Day of embryo transfer (relative to the day of follicle puncture) and number of transferred embryos | 12 months
Luteal phase support (LPS): product, dose and duration of administration | 12 months
User satisfaction with the Ovaleap®-pen | 12 months
  Patient Questionnaire completed by patient
"Baby-Take-Home-Rate" (live-births). | 12 months
Rate of multiple pregnancies (twins, triplets, quadruplets). | 12 months
Frequency and intensity of adverse drug reactions (ADRs) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (37):
- Germany (37):
  - Teva Investigational Site 034, Aalen, Baden-Wurttemberg
  - Teva Investigational Site 033, Kempten (Allgäu), Bavaria
  - Teva Investigational Site 026, München, Bavaria
  - Teva Investigational Site 032, Regensburg, Bavaria
  - Teva Investigational Site 035, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Teva Investigational Site 036, Aalen
  - Teva Investigational Site 004, Berlin
  - Teva Investigational Site 015, Berlin
  - Teva Investigational Site 017, Berlin
  - Teva Investigational Site 027, Berlin
  - Teva Investigational Site 031, Berlin
  - Teva Investigational Site 022, Bielefeld
  - Teva Investigational Site 013, Dortmund
  - Teva Investigational Site 003, Düsseldorf
  - Teva Investigational Site 010, Düsseldorf
  - Teva Investigational Site 011, Essen
  - Teva Investigational Site 025, Esslingen am Neckar
  - Teva Investigational Site 012, Großhansdorf
  - Teva Investigational Site 037, Hamburg
  - Teva Investigational Site 016, Hanover
  - Teva Investigational Site 028, Hildesheim
  - Teva Investigational Site 021, Kiel
  - Teva Investigational Site 029, Leipzig
  - Teva Investigational Site 014, Ludwigsburg
  - Teva Investigational Site 020, Lübeck
  - Teva Investigational Site 023, Magdeburg
  - Teva Investigational Site 006, München
  - Teva Investigational Site 030, München
  - Teva Investigational Site 018, Münster
  - Teva Investigational Site 009, Osnabrück
  - Teva Investigational Site 007, Regensburg
  - Teva Investigational Site 002, Rostock
  - Teva Investigational Site 008, Saarbrücken
  - Teva Investigational Site 019, Stuttgart
  - Teva Investigational Site 005, Ulm
  - Teva Investigational Site 024, Ulm
  - Teva Investigational Site 001, Wiesbaden

REFERENCES:
- [Derived] Sydow P, Gmeinwieser N, Pribbernow K, Keck C, Wiegratz I. Effectiveness and safety of follitropin alfa (Ovaleap(R)) for ovarian stimulation using a GnRH antagonist protocol in real-world clinical practice: a multicenter, prospective, open, non-interventional assisted reproductive technology study. Reprod Biol Endocrinol. 2020 May 26;18(1):54. doi: 10.1186/s12958-020-00610-2. PMID 32456636